CLINICAL TRIAL: NCT06250101
Title: Study 5: Effects of Semantic Support
Brief Title: Training Grammar With Meaning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Elena Plante, Professor, University of Arizona
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLD-Tx2
Record Dates: First submitted 2024-01-23; First posted 2024-02-08 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Language Disorders in Children

STUDY DESIGN:
Intervention Model Description: Hybrid single subject/group design
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Caregivers are not informed of their child's treatment target until after treatment concludes.
  The clinician measuring retention of learning has not treated the children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grammar treatment including semantic support (Experimental): Children receiving grammatical treatment will also receive a simple explanation concerning the meaning of verbs used to elicit grammatical forms.
  Interventions: Behavioral: Enhanced Conversational Recast treatment
- Grammatical treatment excluding semantic support (Active Comparator): Children receiving grammatical treatment will not receive any explanation concerning the meaning of verbs used to elicit grammatical forms.
  Interventions: Behavioral: Enhanced Conversational Recast treatment

INTERVENTIONS:
Behavioral: Enhanced Conversational Recast treatment — In the context of child-friendly activities, the clinician prompts the child to attempt to use the grammatical form targeted in the treatment. The clinician immediately restates the child's attempt (i.e., the recast), correcting any ungrammatical elements. Clinicians elicit and recasts 24 utterances per session.

SUMMARY:
This study will enroll children between the ages of 4 and 6 years of age who exhibit significant difficulty developing language skills without any other handicapping conditions. Children will receive standardized language, hearing, and cognitive testing to confirm a diagnosis of developmental language disorder. Children will be enrolled in a half-day summer camp program for six weeks during which they will receive treatment designed to improve their language skills. Children will be seen again approximately six weeks after the end of treatment to determine how much learning they have retained.

DETAILED DESCRIPTION:
Children between 4 years, 0 months and 6 years 11 months are eligible. A diagnosis of developmental language disorders will be confirmed as normal nonverbal cognitive function, passing a pure-tone audiometric screening, and a test score consistent with developmental language disorder on a standardized language test, and parent report of no other diagnosed handicapping condition. Speech skills and vocabulary skills will be described via standardized testing.

Children enrolled in treatment are seen for up to 28 consecutive weekdays. The study starts with three days of baseline assessment of morpheme use for potential treatment targets. Two are selected for study, with one treated and one tracked over the course of treatment. Treatment is embedded in child-friendly activities like games, book reading, and craft activities. Children are prompted to use the treated morpheme in conversation. Immediately following this attempt, the treating clinician repeats the child's utterance, correcting any ungrammatical forms. Half of the children will also receive explanations of what the key words in sentences mean (e.g., to twirl means to turn around fast). Generalization to untreated contexts is assessed 2-3 times weekly. Retention of learning is measured about six weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

Language scores consistent with a developmental language disorder nonverbal cognitive scores consistent with normal-range intellectual functioning

Exclusion Criteria:

hearing loss Intellectual disability Other handicapping conditions

Ages: 48 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-10-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plante E, Ogilvie T, Vance R, Aguilar JM, Dailey NS, Meyers C, Lieser AM, Burton R. Variability in the language input to children enhances learning in a treatment context. Am J Speech Lang Pathol. 2014 Nov;23(4):530-45. doi: 10.1044/2014_AJSLP-13-0038. PMID 24700145
- [Background] Meyers-Denman CN, Plante E. Dose Schedule and Enhanced Conversational Recast Treatment for Children With Specific Language Impairment. Lang Speech Hear Serv Sch. 2016 Oct 1;47(4):334-346. doi: 10.1044/2016_LSHSS-15-0064. PMID 27701629
- [Background] Plante E, Mettler HM, Tucci A, Vance R. Maximizing Treatment Efficiency in Developmental Language Disorder: Positive Effects in Half the Time. Am J Speech Lang Pathol. 2019 Aug 9;28(3):1233-1247. doi: 10.1044/2019_AJSLP-18-0285. Epub 2019 Jul 25. PMID 31343897
- [Background] Sweeney L, Plante E, Mettler HM, Hall J, Vance R. Less Versus More: The Effect of Recast Length in Treatment of Grammatical Errors. Lang Speech Hear Serv Sch. 2024 Jan 11;55(1):152-165. doi: 10.1044/2023_LSHSS-23-00049. Epub 2023 Dec 1. PMID 38039976

RESULTS

PARTICIPANT FLOW:
Groups:
- Semantic Support: Children are provided a brief definition of the verb they will hear in the recast (i.e., restatement of the child's utterance, correcting ungrammatical portions) prior to clinician administration of the recast.
- No Semantic Support: Children are not provided information on the meaning of the verb they will hear in the recast (i.e., restatement of the child's utterance, correcting ungrammatical portions) prior to clinician administration of the recast.
Period: Overall Study
Arm/Group | Semantic Support | No Semantic Support
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Excessive absenteeism | 1 | 0

BASELINE CHARACTERISTICS:
Population: Children are provided with 10 opportunities on each of 3 consecutive days to use grammatical forms that might be selected for treatment.
Units Other Than Participants: daily use of grammatical forms
Groups:
- Grammatical Treatment Excluding Semantic Support: Children receiving grammatical treatment do not receive any explanation concerning the meaning of verbs used to elicit grammatical forms.
  Enhanced Conversational Recast treatment: In the context of child-friendly activities, the clinician prompts the child to attempt to use the grammatical form targeted in the treatment. The clinician immediately restates the child's attempt (i.e., the recast), correcting any ungrammatical elements. Clinicians elicit and recasts 24 utterances per session.
- Total: Total of all reporting groups
Arm/Group | Grammar Treatment Including Semantic Support | Grammatical Treatment Excluding Semantic Support | Total
Number analyzed (Participants) | 12 | 12 | 24
Number analyzed (daily use of grammatical forms) | 360 | 360 | 720
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4 (.5) | 4 (.5) | 4 (.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One child was withdrawn due to excessive absences.
  Participants
    number analyzed (Participants) | 11 | 12 | 23
    Female | 7 | 9 | 16
    Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 4 | 5 | 9
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Children are provided with 10 opportunities to use grammatical forms each day for three days pretreatment to determine possible treatment targets.
  participants
    United States | 12 | 12 | 24
Average percent use of grammatical forms [Mean (Standard Deviation); unit: Average percent correct use over 3 days] — Average number of times the grammatical form was used correctly, out of 10 opportunities each session, over 3 consecutive sessions. The numbers are expected to be small because grammatical forms chosen for treatment were those rarely if ever used correctly prior to treatment. Population: The values are identical, primarily because we balance the groups for pretreatment use.
  Average percent correct use over 3 days | 6 (4) | 6 (4) | 6 (4)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Use of Treated Grammatical Forms in Untreated Contexts
Description: Clinicians elicit ten uses of the trained grammatical form using toys, activities, and vocabulary with-held from treatment sessions. This is done in a conversational interaction between the clinician and child during play or stories using toys and is referred to as a 'generalization probe'. Because children begin treatment with different levels of pretreatment use, measures like percent use at the end of treatment do not accurately reflect treatment effects. Instead, for each child, data from three generalization probes obtained over a week at the end of treatment are averaged. This average, minus the average of three consecutive pre-treatment probe sessions, divided by the standard deviation of the three end-treatment probes constitutes a Generalization d. This reflects for the amount of change each individual child showed from their pre-treatment baseline, in units of standard deviation. The Generalization d serves as the dependent measure for group statistical analysis.
Time Frame: Three days over the course of the final week (week 5) of treatment
Population: One child was withdrawn from the study due to excessive absentee-ism.
Measure: Mean (Standard Deviation); unit: Generalization d
Arm/Group | Semantic Support | No Semantic Support
Number analyzed (Participants) | 11 | 12
Generalization d | 6.6 (6.9) | 5.8 (7.4)
Statistical Analysis 1: Comparison: Semantic Support vs No Semantic Support; This analysis tests for the overall effectiveness in the study. Groups are collapsed for analysis; Test type: Superiority — We hypothesized a larger change in performance on treated than untreated grammatical forms; Bayesian statistics do not use p values; Bayesian Mann-Whitney U Bayes Factor = 1.06, 1.1% CI 2-sided [.05 to 1.6] — This is the effect size corresponding to a Bayes Factor of 195.4
Statistical Analysis 2: Comparison: Semantic Support vs No Semantic Support; This is a test for differences in the treatment condition (Semantic support vs. No semantic support); Test type: Superiority — We tested for superiority of either condition; Bayesian analyses do not use p values; effect size of Bayes Factor = .05, .02% CI 2-sided [.05 to .07] — This effect size is associated with a Bayes Factor of 2.5

2. Primary Outcome: Change in the Use of Untreated Grammatical Forms in Untreated Contexts
Description: Clinicians elicit ten uses of the trained grammatical form using toys, activities, and vocabulary with-held from treatment sessions. This is done in a conversational interaction between the clinician and child during play or stories using toys and is referred to as a 'generalization probe'. Because children begin treatment with different levels of pretreatment use, measures like percent use at the end of treatment do not accurately reflect treatment effects. Instead, for each child, data from three generalization probes obtained over a week at the end of treatment are averaged. This average, minus the average of three consecutive pre-treatment probe sessions, divided by the standard deviation of the three end-treatment probes constitutes a Generalization d. This reflects the amount of change each individual child showed from their pre-treatment baseline, in units of standard deviation. The Generalization d serves as the dependent measure for group statistical analysis.
Time Frame: Three days over the course of the final week (week 5) of treatment
Population: One child was withdrawn due to excessive absenteeism.
Measure: Mean (Standard Deviation); unit: Generalization d
Arm/Group | Semantic Support | No Semantic Support
Number analyzed (Participants) | 11 | 12
Generalization d | .02 (4.1) | .03 (5.6)
Statistical Analysis 1: Comparison: Semantic Support vs No Semantic Support; This tests to determine whether untreated grammatical forms changed over the period of treatment; Test type: Equivalence — 1/BF is used to test for equivalence of two conditions; Bayesian analysis does not use p values; effect size of Bayes Factor = 0.03, -.03% CI 2-sided [-.4 to .4] — This effect is associate with a Bayes factor 0f 4.4

3. Primary Outcome: Retention of Trained Grammatical Forms
Description: Clinicians elicit ten uses of the trained grammatical form using toys, activities, and vocabulary with-held from treatment sessions. This is done in a conversational interaction between the clinician and child during play or stories using toys and is referred to as a 'retention probe' when done, as here, after a period of no treatment. The dependent measure is the number correct out of 10 opportunities for use of the grammatical form.
Time Frame: 1 day, 1-2 months after the end of treatment
Population: The analysis compares the mean performance at the end of treatment (3 data points) to retention performance 1-2 months post treatment (1 data point). One child was withdrawn due to excessive absenteeism.
Measure: Mean (Standard Deviation); unit: percentage of correct use
Arm/Group | Semantic Support | No Semantic Support
Number analyzed (Participants) | 11 | 12
percentage of correct use | 2.1 (3.5) | 4.6 (3.2)
Statistical Analysis 1: Comparison: Semantic Support vs No Semantic Support; This analysis tests for differences between the two condition for retention of trained grammatical forms over time; Test type: Superiority — We tested for superiority of either condition; Bayesian statistics do not use p values; effect size of Bayes Factor = .06, 1.3% CI 2-sided [-.1 to 1.5] — This effect size is associated with a Bayes Factor of 1.4

4. Primary Outcome: Retention of Untrained Grammatical Forms
Description: as for outcome 3
Time Frame: 1 day, 1-2 months from the end of treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of correct use
Arm/Group | Semantic Support | No Semantic Support
Number analyzed (Participants) | 11 | 12
Percentage of correct use | 1.4 (2.7) | 1.3 (2.7)
Statistical Analysis 1: Comparison: Semantic Support vs No Semantic Support; Test for retention of untreated grammatical forms after a period of no treatment; Test type: Equivalence — 1/BF tests for equivalence; Bayesian analyses do not use p values; effect size of Bayes Factor = .3, .4% CI 2-sided [-.1 to .7] — This is associated with a Bayes Factor of 1.5

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Semantic Support | No Semantic Support
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT06250101/Prot_SAP_000.pdf